CLINICAL TRIAL: NCT05026814
Title: Clitoral Reconstruction (CR) in FGM/C Patients: Assessment of Multidisciplinary Care
Brief Title: Clitoral Reconstruction (CR) in FGM/C Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01190; bb21Sartorius
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Female Genital Mutilation / Cutting (FGM/C)
Keywords: Clitoral Reconstruction (CR); Psychosexual care (PC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with FGM/C: Women who requested clitoral reconstruction after FGM/C between 01/2013 until 04/2021 and underwent multidisciplinary care consisting of psychosexual care (PC) with or without CR. To be included the women had to attend at least one session with the psychologist as part of psychosexual care.
  Interventions: Other: Interview after one year or more from the treatment received

INTERVENTIONS:
Other: Interview after one year or more from the treatment received — Questionnaires to evaluate the satisfaction with treatment, the motivations and expectations for the treatment, the general well-being, the sexual function and the genital selfimage

SUMMARY:
Surgical interventions to reconstruct the vulva together with psychosexual care have been proposed as a multidisciplinary care concept for women who have undergone female genital mutilation/cutting (FGM/C).

This cross-sectional study is to assess the experiences of multidisciplinary care of women who request CR at Geneva University Hospital (HUG) in order to analyze the expectations and motivations for clitoral reconstruction, to study the reasons for deciding against or in favor of CR and to study the outcome of the care received (CR+ psychosexual care versus psychosexual care alone) in sexual response, eventual dyspareunia, genital self-image and overall satisfaction through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent of the present study
* French and / or English speaking

Exclusion Criteria:

* Insufficient knowledge of project language (French/English)
* No informed consent
* Inability to sign consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: FGM/C patients of the FGM/C outpatient clinic of HUG within the time frame of 01/2013 until 04/2021
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
General satisfaction with multidisciplinary care | one time assessment at baseline
  General satisfaction with multidisciplinary care rated on a scale from 0 to 10 (0=totally unsatisfied, 10: totally satisfied)

SECONDARY OUTCOMES:
General satisfaction with subdomain CR and psychosexual care | one time assessment at baseline
  General satisfaction with subdomain CR and psychosexual care rated on a scale from 0 to 10 (0=totally unsatisfied, 10: totally satisfied)
General satisfaction with subdomain CR alone | one time assessment at baseline
  General satisfaction with subdomain CR alone rated on a scale from 0 to 10 (0=totally unsatisfied, 10: totally satisfied)
General satisfaction with subdomain psychosexual care | one time assessment at baseline
  General satisfaction with subdomain psychosexual care rated on a scale from 0 to 10 (0=totally unsatisfied, 10: totally satisfied)
General satisfaction after CR with sexual response | one time assessment at baseline
  General satisfaction after CR with sexual rated on a scale from 0 to 10 (0=totally unsatisfied, 10: totally satisfied)
General satisfaction after CR with genital image | one time assessment at baseline
  General satisfaction after CR with genital rated on a scale from 0 to 10 (0=totally unsatisfied, 10: totally satisfied)
General satisfaction after CR with pain | one time assessment at baseline
  General satisfaction after CR with pain rated on a scale from 0 to 10 (0=totally unsatisfied, 10: totally satisfied)
General satisfaction after CR with female identity | one time assessment at baseline
  General satisfaction after CR with female identity rated on a scale from 0 to 10 (0=totally unsatisfied, 10: totally satisfied)
Female Genital Self Image Scale (FGSIS) | one time assessment at baseline
  The FGSIS is a measurement instrument consisting of seven items to assess female genital self-image. The questions relate to women's feelings and beliefs about their own genitals. A total score is calculated using a four-point response scale (strongly agree, agree, disagree, and strongly disagree).
World Health Organization (WHO)-Five Well-Being Index | one time assessment at baseline
  The WHO-Five Well-Being Index is a questionnaire consisting of five questions to assess wellbeing. For each question, scores from 0 to 5 can be given. By adding up the values for the answers, a total value is obtained, whereby a low total value corresponds to low well-being

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Abdulcadir, PD Dr. med., Principal Investigator — Department of Obstetrics and Gynecology, University Hospital of Geneva (HUG)
Locations (1):
- University Hospital of Geneva (HUG), Department of Obstetrics and Gynecology, Geneva, Switzerland

REFERENCES:
- [Derived] Meyer M, Sartorius G, Abdulcadir J. Clitoral reconstruction and psychosexual care after female genital mutilation/cutting: Assessment of multidisciplinary care. Womens Health (Lond). 2025 Jan-Dec;21:17455057251315814. doi: 10.1177/17455057251315814. Epub 2025 Mar 31. PMID 40162955